CLINICAL TRIAL: NCT00229567
Title: A Randomised Controlled Trial of Lidocaine Infusion Plus Ketamine Injection Versus Placebo to Decrease Postoperative Ileus
Brief Title: Intra-op Lidocaine and Ketamine Effect on Postoperative Bowel Function
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: insufficient numbers of eligible patients as laparscopic surgery increased and open surgery decreased.
Sponsor: University of Saskatchewan (Other)
Collaborators: Saskatoon Health Region (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Bio-REB 03-1316
Record Dates: First submitted 2005-09-27; First posted 2005-09-29 (Estimated); Last update posted 2007-04-19 (Estimated); Status verified 2007-04

CONDITIONS: Colorectal Cancer
Keywords: ketamine; lidocaine; postoperative ileus; randomized controlled trial; acute postoperative pain
MeSH Terms: conditions — Colorectal Neoplasms; Pain, Postoperative | interventions — Ketamine

INTERVENTIONS:
Drug: Lidocaine infusion plus ketamine injection

SUMMARY:
Bowel function after bowel surgery is delayed (postoperative ileus)by both opiates and the surgery itself. We hypothesized that decreasing opiate use by other analgesics will speed the return of bowel function after surgery. Lidocaine and Ketamine are drugs that appear to be synergistic and do not slow peristalsis. This study is a Randomised Controlled Trial of Lidocaine Infusion Plus Ketamine Injection versus Placebo to to determine whether they will decrease opiate use and then whether decreased opiate use will speed the return of bowel function.

DETAILED DESCRIPTION:
Introduction: Postoperative ileus is a normal response to the surgical handling of bowel that causes transient impairment of bowel motility after abdominal surgery. It is characterized by distension, absence of bowel sounds, and lack of passage of flatus and stool. The duration of postoperative ileus is related to the degree of surgical manipulation and the location of surgery. Colonic surgery is associated with the longest duration of ileus. Morphine patient-controlled intravenous analgesia (PCIA) is commonly used to provide pain control after bowel surgery. The bowel wall contains opiate receptors that decrease bowel peristalsis in the presence of morphine. Thus, both surgery and PCIA slow return of normal bowel function.

Lidocaine and ketamine are non-opioid analgesics that have been shown to be safe and efficacious in low doses when combined with morphine for post-operative pain control. Since the addition of lidocaine or ketamine to a morphine PCIA regimen results in lower total use of morphine, and since lidocaine or ketamine does not slow peristalsis, , it is reasonable to expect that low-dose lidocaine or ketamine plus PCIA morphine will result in faster return of bowel function than PCIA morphine alone.

Intravenous lidocaine was first shown to relieve cancer pain in the 1950s. Since then, intravenous lidocaine has been shown also to relieve pain after a wide variety of surgeries. Ketamine is a non-opioid analgesic that has been shown to be safe and efficacious in very low doses when combined with morphine for post-operative pain control . A review of ketamine for postoperative pain control recently completed by Dr McKay has shown that ketamine is most efficacious when given after a painful surgical insult, and that preoperative bezodiazepines prevent ketamine-induced hallucinations (submitted for publication). Groudine, in patients undergoing radical retropubic prostatectomy, determined that intravenous lidocaine infusion intraoperatively decreased the duration of postoperative ileus, decreased the pain scores postoperatively, and resulted in a 50% reduction in morphine use, and a 20% reduction in hospitalization time. This was felt to be due to early ambulation, earlier times to passing gas and having a bowel movement, and faster advancement to a full diet and oral analgesics. Lidocaine plasma levels were well below toxic range.

We propose a double-blind placebo-controlled study of patients undergoing elective or urgent colon surgery with an anastomotic procedure. All patients will receive normal PCA morphine in addition to study drugs or placebo. Research will be conducted at Saskatoon teaching hospitals. This procedure was chosen as it is associated with a longer duration of ileus compared to other abdominal surgeries and more likely to show a significant treatment effect.

If previous data is applicable to colonic surgery then we can expect a decrease in postoperative analgesic requirements, earlier return of bowel function, earlier progression to full diet and earlier discharge dates.

The dose of lidocaine we propose has been shown to be safe in thousands of patients for whom it was used to treat arrhythmias; that of ketamine in more than twenty studies of postoperative pain control.

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 79
* booked for urgent or elective colon surgery undergoing a left, right, or transverse hemicolectomy via laparotomy

Exclusion Criteria:

* patients requiring emergency surgery
* pregnant subjects or those who might be pregnant
* subjects allergic to lidocaine, ketamine, morphine, naproxen, or acetaminophen
* subjects with epidural analgesia
* subjects unable to understand and implement a Patient-Controlled Intravenous Analgesia system
* subjects who do not know English well enough to understand the consent form and assessments
* subjects with known hepatic or renal failure or cardiac dysrhythmias or atrioventricular block
* patients with pre-existing functional bowel motility disorders including Crohn's disease and ulcerative colitis
* daily use of laxatives, inability to have a bowel movement without laxatives, use of suppositories or enemas on a daily basis, or use of antimotility agents
* patients with Parkinson's disease

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2005-09; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Mean time after surgery to completion of the following postoperative markers:
drinking and retaining 500ml clear fluids,
presence of bowel sounds
passage of flatus, and
passage of stool.

SECONDARY OUTCOMES:
pain after cough by VAS
narcotic usage
nausea
vomiting
infection, dehiscence and other surgical complications
time to readiness for discharge from hospital

CONTACTS AND LOCATIONS:
Overall Officials: William PS McKay, MD, Principal Investigator — University of Saskatchewan
Locations (1):
- Saskatoon Health Region, 410 22nd Street East, Saskatoon, Saskatchewan, Canada